CLINICAL TRIAL: NCT00589095
Title: Early Detection of Glioblastoma Multiforme (GBM) Treatment Responses Using Multiple Magnetic Resonance Modalities
Status: Terminated | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 0606001531
Record Dates: First submitted 2008-01-02; First posted 2008-01-09 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — gadodiamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: dynamic contrast enhanced magnetic resonance imaging

INTERVENTIONS:
Other: dynamic contrast enhanced magnetic resonance imaging — dynamic contrast enhanced MRI using contrast agent gadodiamide
  Other Names: Omniscan

SUMMARY:
The purpose of this study is to determine whether dynamic contrast enhanced MRI (DCE MRI) and high diffusion weighting MRI may be used to distinguish between favorable and unfavorable responses to therapy of glioblastoma multiforme. Imaging data will be correlated with histopathologic findings and clinical responses to radiation therapy with or without chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* The presence of a primary brain tumor that cannot be completely resected that requires radiation therapy with or without chemotherapy.

Exclusion Criteria:

* Patients who do not have a primary brain tumor or who are unable to tolerate the environment of the MRI scanner

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Yale Brain Tumor Center for management of glioblastome multiforme
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2006-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To detect the early "local" treatment responses from the physician recognized GBM "gross tumor volume" (GTV) | Upon completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Knisely, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States